CLINICAL TRIAL: NCT06668766
Title: Superior Ultrasound-Guided Venous Access: Single-Lumen Midline Catheters vs Long Peripheral IVs for Difficult IV Access in the Emergency Department, A Randomized Controlled Trial
Brief Title: Single Lumen Midline Catheter vs Long Peripheral Intravenous Cather for Difficult Intravenous Access in the ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Alexander Bracey, MD, Associate Research Director, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6890
Record Dates: First submitted 2024-10-17; First posted 2024-10-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Difficult Intravenous Access; Midline Catheter; Peripheral Intravenous Catheter; Emergency Department Patient
Keywords: midline catheter; difficult intravenous access; difficult IV access; USGIV; long peripheral IV; peripheral IV; peripheral intravenous catheter; Emergency department; emergency medicine; single lumen midline catheter; long peripheral intravenous catheter
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: This is a single center, prospective, 2-arm, nonblinded, randomized clinical trial to determine if midline catheters (10 cm) are superior to the long peripheral intravenous catheterss (4.78-cm) may with respect to dwell time, dislodgement and infiltration rates, and patient preference.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 4.78 cm Long Peripheral Intravenous Catheter (Active Comparator): The BD Insyte Autoguard 4.78 cm 18- or 20-gauge needle with self-retraction is currently approved for use by the FDA and by Albany Medical center. The long PIV will be placed using standard aseptic technique (e.g., chlorhexidine prep, sterile gloves, sterile ultrasound probe cover and gel). Once the target vessel is identified, an ultrasound image of the vessel will be captured and recorded with the subject's study ID number in the comments section of the QPATH worksheet to allow for vessel depth and size measurement. Operators will be instructed to use standard techniques in US-guided vascular access.
  Interventions: Device: 4.78 cm Long Peripheral Intravenous Catheter
- 10 cm Single Lumen Midline Catheter (Experimental): The BD Powerglide Pro Midline catheter is currently approved for use by the FDA and by Albany Medical Center. This 18-gauge or 20-guage MC is distinct in that it is a standard 10-cm, does not require premeasurement or trimming of the catheter prior to placement, and features an accelerated Seldinger technique, meaning that it has a built-in deployable internal wire system. Additionally, because it is only 10-cm, it does not require a confirmatory chest x-ray prior to use. The provider will use standard aseptic technique for placing the MC (e.g., chlorhexidine prep, sterile probe cover and gel). Once the target vessel is identified, an ultrasound image of the vessel will be captured and recorded with the subject's study ID number from the randomization packet to allow for vessel depth and size measurement.
  Interventions: Device: 10-cm Single Lumen Mildine

INTERVENTIONS:
Device: 10-cm Single Lumen Mildine — Arm Description: The BD Powerglide Pro Midline catheter is currently approved for use by the FDA and by Albany Medical Center. This 18-gauge or 20-guage MC is distinct in that it is a standard 10-cm, does not require premeasurement or trimming of the catheter prior to placement, and features an accelerated Seldinger technique, meaning that it has a built-in deployable internal wire system. Additionally, because it is only 10-cm, it does not require a confirmatory chest x-ray prior to use. The provider will use standard aseptic technique for placing the MC (e.g., chlorhexidine prep, sterile probe cover and gel). Once the target vessel is identified, an ultrasound image of the vessel will be captured and recorded with the subject's study ID number from the randomization packet to allow for vessel depth and size measurement.
  Arms: 10 cm Single Lumen Midline Catheter
Device: 4.78 cm Long Peripheral Intravenous Catheter — The BD Insyte Autoguard 4.78 cm 18- or 20-gauge needle with self-retraction is currently approved for use by the FDA and by Albany Medical center. The long PIV will be placed using standard aseptic technique (e.g., chlorhexidine prep, sterile gloves, sterile ultrasound probe cover and gel). Once the target vessel is identified, an ultrasound image of the vessel will be captured and recorded with the subject's study ID number in the comments section of the QPATH worksheet to allow for vessel depth and size measurement. Operators will be instructed to use standard techniques in US-guided vascular access.
  Arms: 4.78 cm Long Peripheral Intravenous Catheter

SUMMARY:
Many patients in the emergency department have veins that are difficult to get an intrevenous (IV) catheter into (called "difficult IV access"). These patients may require other methods to obtain access to a vein for administration of the necessary medications. The 2-inch long IV is most commonly used in emergency departments for people with difficulty IV access. Typically, a healthcare worker will use an ultrasound to help to see the veins underneath the skin while inserting the IV into the vein. That is, the ultrasound helps the healthcare worker visualize veins that are deeper in the arm and may not be felt through the skin. Another device that can be used is a 4-inch midline catheter. This device is less commonly used as many emergency departments do not have participants available, but it serves the same purpose as the 2-inch long IVs (that is, to give medicine into the vein and sometimes to take blood). A 4-inch midline catheter is similar to a 2-inch long IV, but has a few differences. First, the 4-inch midline catheter is even longer than the 2-inch long IV. The 4-inch midline catheter is 10-cm (about 4-inches or the size of 4 quarters side-by-side), while the 2-inch long IV is 4.78-cm (nearly 2-inches or two quarters side-by-side). Second, the 4-inch midline catheter is inserted into using a guidewire to help move the catheter in the vein (similar in concept to a train moving along a track), while the 2-inch long IV does not have this guidewire. The guidewire does not hurt and most do not know it is being used. It is just an additional step to help guide the catheter in the vein. The investigators are conducting this research study to determine which catheter is better for patients with difficult IV access: the 4-inch midline catheter or the 2-inch long IV.

DETAILED DESCRIPTION:
Intravenous (IV) access is among the most commonly performed procedures performed in the acute care setting. IV access is also essential for the delivery critical care in the emergency department (ED) setting, as it allows for the collection of blood samples that can be sent for serum laboratory studies and the administration of medications, several of which are potentially lifesaving. While this procedure is common, achieving IV access may be challenging with prior work demonstrating that 1 in 9 patients may be considered to have difficult IV access in the ED setting. These patients may have delays in delivery of care leading to potential increased risk of morbidity and mortality.

There are many vascular access devices (VADs), each of which has different characteristics. For example, traditional IVs are typically 3-cm in length, while "long" and "ultralong" IVs are 4.78-cm and 6.35-cm respectively, with shorter catheters most often reserved for landmark based peripheral IV (PIV) placement while longer PIVs are used for deeper vessels with US guidance. It has been demonstrated that shorter IV catheters placed in deeper vessels under ultrasound (US) guidance have significantly shorter dwell times (duration before failure) than those with longer catheter length. One study demonstrated an IV failure rate of 8% within the first hour when using long 4.78-cm IV for deep vessels under US guidance. Another study of patients undergoing US guided IV insertion with an "ultralong" 6.35-cm PIV catheter versus "standard long" 4.78-cm PIV reported a median dwell time of 136 hours and 96 hours respectively. Furthermore, 12-cm PIVs inserted using Seldinger technique have been shown to have a longer mean dwell time. Another study demonstrated a mean dwell time of 6.2 days in 12-cm, US-guided, Seldinger-technique PIVs compared to the 3.5 days with a 5 cm, US-guided, non-Seldinger-technique PIV. Therefore, it is reasonable to assume that catheter length has a direct influence on catheter dwell time.

An especially promising area of longer IVs is in the administration of medications that are used to artificially elevate blood pressure (e.g., vasopressors). Traditionally such medications are administered through central venous access via a central venous catheter (CVC). This practice was born out of fear of vasopressor extravasation from peripheral administration that could result in tissue necrosis and/or limb ischemia. Such reports, however, are based on older case reports while recent robust literature indicates that such events are fleetingly rare.

There is burgeoning literature supporting the use of midline catheters (MCs) for those patients requiring intermediate duration of IV access and who may have difficult IV access. MCs are a heterogenous group of VADs that may be single or dual lumen and may feature fixed or trimmable catheters. MCs are almost exclusively placed using ultrasound guidance and can be placed rapidly as many feature quick or accelerated Seldinger technique (i.e., needle into vein, wire through needle, needle removed, catheter over wire, and finally wire removed with all steps occurring within a single device). Seldinger technique is a widely established technique for IV catheters inserted into the central venous system and may confer benefit when accessing peripheral veins as well.

MCs may have advantages over PIVs for the management of critically ill patients in the ED setting for at least three reasons. First, despite the heterogeneity in length, gauge, and insertion technique, MCs are categorically more reliable than PIVs with existing studies showing average dwell times of 16.3 days for MC versus 4.8 days for PIVs. Second, MCs can serve as long term vascular access, with one study demonstrating that 68% of patients who underwent MC placement never required additional IV insertion through the remainder of their hospitalization. Third, some MCs are capable of providing multiple ports of access at a single site, which is helpful when needing to infuse several medications simultaneously as is common in the management of critically ill patients.

While it has been demonstrated that increasing PIV catheter lengths are associated with increased duration of PIV dwell times, it is not known whether MCs confer benefit, such as increased dwell time, over long PIVs. In addition, there is at least the perception MCs take longer to place than PIVs. Finally, it is largely unknown whether patient or provider preferences differ for each type of line. Therefore, in order to answer these questions, the investigators intend to perform a randomized clinical trial of ultrasound-guided long PIVs versus ultrasound-guided MCs in the ED patients with difficult IV access.

Importantly, both ultrasound-guided MCs and ultrasound-guided PIVs are approved for standard of care (SOC) use at Albany Medical Center (AMC) for patient care.

Specific Aims

Aim 1: To determine if US-guided MCs (10-cm) have longer dwell times (a longer duration before failure) than US-guided long PIVs (4.78-cm).

There are several reasons why long PIVs may fail. Long PIVs (4.78-cm) are shorter than MCs (10 cm), and shorter catheters may fail due to dislodgement out of the vein which can be a result of malposition as well as displacement during routine clinical course. Other common reasons for failure include pain, infiltration (i.e., when fluid leaks into the surrounding tissues rather than entering the blood stream), device leakage, device kinking, catheter occlusion, or phlebitis (i.e., painful inflammation after IV insertion). The investigators suspect that longer MCs (10-cm) placed with a guidewire (i.e., Seldinger technique) will confer benefit in the form of increased catheter dwell time and thus lower rates of failure when compared to long PIVs (4.78-cm).

Aim 2: To compare the complication rates of MCs (10-cm) versus long PIVs (4.78-cm) in ED patients with difficult IV access.

This is an exploratory analysis aimed at investigating complication rates of MCs vs long PIVs. Complications include but are not limited to the following: displacement, extravasation, arterial puncture, infection, deep vein thrombus, failure to aspirate, and multiple IV insertion attempts.

Aim 3: To determine patient experience, satisfaction, and preference; provider perceptions and cognitive load; and operational characteristics for each device placement.

Patient experience as measured by pain score, satisfaction, and preference will be determined based on an administered survey. The investigators theorize that a higher failure rate of long PIVs (4.78-cm) may lead to additional needle sticks for re-catheterization, resulting in patients preferring the more durable midline catheter to avoid additional needle sticks despite MC (10-cm) placement being marginally more invasive. Provider cognitive load and time to placement will be measured by a provider questionnaire and time-motion analysis. The investigators theorize that the cognitive load and time to placement will be equivalent in both arms. In addition, the investigators will record operational characteristics of the device placement and use including the number of catheters used for vascular access attempts, the time required for placement of each device, vascular access used for CT scanning, vascular access used for vasopressor administration, need for additional IV access during ED visit (MC, PIV, or central venous catheter (CVC)), catheter occlusion, and need for additional IVs during hospitalization. The investigators will also record patient arm circumference, and catheter length within the vessel to determine if these factors influence catheter dwell time.

This is a single center, prospective, 2-arm, nonblinded, randomized clinical trial to determine if MCs (10 cm) are superior to the long PIVs (4.78-cm) with respect to dwell time, dislodgement and infiltration rates, and patient preference. This study will be entered into clinicaltrials.gov.

Approval of this protocol from other departments is unnecessary because (a) the interventions of the study will be done in the ED setting [with only observations of study participants being done on the medical and surgical floors] and (b) all interventions are considered standard of care. Moreover, nursing research committee approval is not necessary because (a) all study procedures will be done by study personnel, (b) all interventions are considered standard of care, and (c) and nurses will not be asked to perform any additional tasks.

Randomization

Prior to the initiation of the study, the investigators will use an online randomizer to create a set of integers, 1 or 2.

https://ctrandomization.cancer.gov/tool/

"1" will be considered "long PIV" while "2" will be considered "single lumen midline catheter." The investigators will generate enough for twice the sample size (see below) with 30 extra to account for possible withdrawal or incomplete data, totaling 270 numbers generated. The investigators will then print these numbers along with the description (i.e., Long PIV or Single lumen midline catheter) on an individual sheet of paper which will be folded and then inserted into opaque envelopes that will then be sealed and only opened after written informed consent has been signed.. These envelopes will be stored under lock and key in the research office in the order in which randomization occurred.

Only after determining eligibility and obtaining consent will research personnel open the next consecutively numbered envelope, taking from the top of the stack. In this way, randomization to either long PIV or single lumen midline catheter will occur in a 1:1 ratio.

Study Devices

Four possible catheters will be used in this comparison: standard long 18- or 20- gauge BD Insyte Autoguard 4.78-cm IV catheters and single lumen 18- or 20-gauge BD Powerglide 10-cm midline catheter. Only 2 different lengths of catheters will be studied, each of which has two different gauge sizes (i.e., circumference). Gauge size will be determined by clinician preference which has no influence on medication administration. Both interventions are considered standard of care in our ED. Device insertion will be performed in the AMC ED. The study devices will be prepared in equipment bundles as below:

Note. While the study devices are long PIVs (4.78-cm) and MCs (10-cm); in the informed consent, the investigators will call these 2 inch and 4 inch for better understanding from the participants.

Equipment Bundles

Pre-prepared bundles will be available following randomization. These kits will be created by the research staff and kept in the research office. Kits will be composed of:

Long PIV Bundle:

* 18-gauge 4.78 cm BD Insyte Autoguard x1
* 20-gauge 4.78 cm BD Insyte Autoguard x1
* Sterile probe cover x1
* Sterile gel packet x1
* J-loop tubing x1
* Saline flush x1
* Sorbaview® transparent dressing and securement device x1
* Chlorhexidine swab x1

MC Bundle:

* 18-gauge 10 cm BD Powerglide Midline Catheter x1
* 20-guage 10 cm BD Powerglide Midline Catheter x1
* Sterile probe cover x1
* Sterile gel packet x1
* J-loop tubing x1
* Saline flush x1
* Statlock® securement device x1
* Transparent dressing x1
* Chlorhexidine swab x1

Study Arms

Patients who sign written informed consent will be randomized into one of two arms: long PIVs or single lumen MCs. Qualified proceduralists (Registered Nurses [RNs], Advanced Practice Provider [APPs], or physicians, all of whom are study team members) who have undergone formal training will perform device insertion in the AMC ED following randomization. MCs and long PIVs are both approved for use and stocked in the AMC ED.

Long PIV arm The BD Insyte Autoguard 4.78 cm 18- or 20-gauge needle with self-retraction is currently approved for use by the FDA and by Albany Medical center. The long PIV will be placed using standard aseptic technique (e.g., chlorhexidine prep, sterile gloves, sterile ultrasound probe cover and gel). Once the target vessel is identified, an ultrasound image of the vessel will be captured and recorded with the subject's study ID number in the comments section of the QPATH worksheet to allow for vessel depth and size measurement. Operators will be instructed to use standard techniques in US-guided vascular access. This includes attempting placement with short-axis out-of-plane technique, visualizing the "vanishing target sign," and confirming catheter placement once deployed with long-axis in-plane view. The amount of catheter in the vessel will be recorded on long access view and calculated by subtracting the total length of the catheter by the amount of catheter external to the vessel by US imaging in the long access. US images will be stored on the QPATH system. Once successful long PIV access has been achieved, a J-loop IV extension tubing will be attached. If needed, blood samples will be drawn at this time. Flushing of the line with sterile saline will then be performed and the J-loop tubing will be clamped to prevent backflow of blood. The catheter will be secured using Sorbaview® transparent dressing and a securement device.

Midline Cather arm The BD Powerglide Pro Midline catheter is currently approved for use by the FDA and by Albany Medical Center. This 18-gauge or 20-guage MC is distinct in that it is a standard 10-cm, does not require premeasurement or trimming of the catheter prior to placement, and features an accelerated Seldinger technique, meaning that it has a built-in deployable internal wire system. Additionally, because it is only 10-cm, it does not require a confirmatory chest x-ray prior to use. The provider will use standard aseptic technique for placing the MC (e.g., chlorhexidine prep, sterile probe cover and gel). Once the target vessel is identified, an ultrasound image of the vessel will be captured and recorded with the subject's study ID number from the randomization packet to allow for vessel depth and size measurement. The vessel will then be selected, and the needle will be guided by ultrasound until venous flash is obtained. The built-in guidewire will be advanced through the needle, and the catheter will be placed over the guidewire via the accelerated-Seldinger technique. The catheter placement will then be confirmed with a long axis view of the catheter in the vessel. The catheter will then be secured in place, and a Tegaderm will be placed over the entire MC insertion site to prevent infection. US imaging confirmation of the catheter in vessel will be stored on the QPATH system. Once successful long PIV access has been achieved, a J-loop IV extension tubing will be attached. If needed, blood samples will be drawn at this time. Flushing of the line with sterile saline will then be performed and the J-loop tubing will be clamped to prevent backflow of blood. The catheter will be secured using Statlock® securement device with a transparent dressing applied over this. A label indicating "Midline Catheter" will be placed on top of the transparent dressing.

QPATH images:

The research personnel performing the IV insertion procedure will save an image of the target vessel on the QPATH storage device. This is a password protected US image storage system that is used in routine clinical care at AMC currently. Research personnel will retrospectively record the depth of the vessel from the skin to the center of the vessel, along with the diameter of the vessel from outer wall to outer wall.

Study Personnel Study personnel will include (a) the proceduralists (qualifications listed below) and (b) the research coordinators. All study personnel will be trained on the informed consent process.

Proceduralists

Proceduralists are study personnel (team members) who are clinicians and have the following qualifications:

1. At least 1-year of experience inserting PIVs with real-time ultrasound guidance
2. Have attended a 1-hour training session with the IV access team at AMC which will include a lecture on technique and a practical session using both long PIVs and MCs
3. Have appropriate clinical credentials (e.g., AMC RN, APP, Resident Physician, Fellow, or Attending Physician)

Proceduralists will also be trained in enrollment, consent, and data collection; and, therefore, will be able to conduct the study in the absence of research coordinator availability (e.g., overnights).

Research Coordinator Research coordinators will be trained in study conduct and supervised by the study investigators. Research coordinators will, when available, obtain informed consent, gather study materials, collect time-motion data, survey providers, survey subjects, perform observations of the IV site, perform chart review, and contact participant by phone when needed.

Study Procedure

Each subject will remain in the study for 1-month following study VAD removal.

The only study intervention visit will be the ED visit and its associated hospitalization. Patients presenting to the AMC ED will be screened for difficult IV access by study personnel by EMR or by referral from clinical staff. Potential study candidates will be approached in the ED by study personnel to assess for eligibility and, if eligible, attempt to obtain informed consent. Research personnel may also include members of the clinical team. If written informed consent is obtained, the subject will be randomized by opening the next consecutively numbered, sealed, opaque envelope containing the arm of the study in which the patient will be enrolled. Study personnel (study team members) will then obtain the appropriate equipment bundle (see above) for the study arm, which will then be given to the clinician who will be performing the procedure.

The proceduralist will apply a tourniquet to either upper extremity (if both are available) and use the ultrasound to identify a target vessel. Both PIVs and MCs can access the veins of the forearm and upper arm. The choice of the size of the VAD gauge (e.g. circumference size) will be at the discretion of the proceduralist. Once a target vessel has been identified, the skin at the anticipated puncture site should be cleansed with the Chlorhexidine swab. After cleansing, the VAD will be inserted into the vessel. Confirmation of successful VAD placement should be performed by viewing the vein in both short and long axis views with the US. These images will be saved into the QPATH system. Following confirmation of placement, a J-loop IV extension that has been pre-flushed with saline will be attached to the VAD and flushed again with sterile saline. Long PIVs should be secured with the Statlock® device followed by transparent dressing if using MC or with the Sorbaview® transparent dressing and securement device if using the long PIV.

Once subjects go up to the inpatient floor, the managing clinical team will manage the subject at their discretion. This may include, for example, placing a MC in a patient randomized to long IV and vice versa. The decision to continue use or remove study devices will be at the discretion of the clinical team and subjects may withdraw from the study at any time and may request for their VAD to be removed. The device will be removed per usual clinical care, which is typically with a long IV by a patient's nurse or patient care technician, and with a MC by a patient's nurse or provider. Per AMC hospital "Policy and Procedure 23: Recommendations for the Prevention of Nosocomial Intravascular Device Related Infections" page 2, PIVs must be removed and replaced "only when clinically indicated" while MCs must be removed and replaced "only when there is a specific indication or as per manufacturer instructions."

If the proceduralist cannot successfully insert a catheter, then this procedure will be aborted, and the clinical staff will be alerted of this. This will be recorded in the notes of the data collection section. The clinical staff would then be responsible for obtaining IV access, as is routine clinical care.

Data collection Prior to subject enrollment, study personnel will screen potential subjects and record demographic data in a screening log. The screening log will include all subjects that are approached and screened for eligibility in the study and will serve to ensure that the investigators have adequate reporting of subjects that are screened and reasons for exclusion in this study. Furthermore, the investigators would like to collect basic demographic data on those not included in the study. Specifically, the investigators intend to collect MRN, age, race, and sex. The purpose for including these data is to be able to report that the investigators are able to report whether there is a discrepancy in those included in the study vs those that were screened out. The investigators have included the screening form that the investigators intend to collect. This screening form will be kept in a password protected folder in the study Microsoft Teams folder.

Data will be collected directly from the subject, the medical record (EHR), and/or through direct observations. Data will be collected in paper records and then transcribed into RedCap or directly into entered into REDCap™, as well as an enrollment log stored on the hospital departmental drive, which will be password protected and stored on the AMC Teams folder. Data recorded on paper sheets (and consent forms) will be stored in locked filing cabinets in the Emergency Medicine administrative offices which only the research coordinator and the PI can access.

When the research coordinator is available, the research coordinator will perform the time-motion measurements using a stopwatch. [Note, the research coordinator may not be available for every patient recruited and enrolled. For example, during overnights, the principal investigator may enroll a patient without the research coordinator. In these circumstances the investigators will not be able to capture the time motion portion of the data. Nevertheless, the time motion data still have some validity, as the randomization will occur after the study personnel are aware of whether the time motion data will be collected. In this way, the subjects on whom the investigators collect time motion data will be equally randomized to each study arm.]

The research personnel performing the IV insertion procedure will save an image of the target vessel on the QPATH storage device. This is a password protected US image storage system that is used in routine clinical care at AMC currently. Research personnel will retrospectively record the depth of the vessel from the skin to the center of the vessel, along with the diameter of the vessel from outer wall to outer wall.

Following placing the VAD and securing the line, study personnel will measure the subject's upper and lower arm circumference midway between the shoulder and elbow and elbow and wrist respectively using a tape measure and record this information.

After the procedure and physical measurements are complete, study personnel will administer a questionnaire to the subject about their experience with the insertion of the VAD and will administer a questionnaire to the proceduralist regarding their cognitive load. When a research associate is not available and the proceduralist is acting in the role of data collection as well, the proceduralist will slef-administer the survey. (Please, see Data Elements in the appendix.) Subject contact information including phone number (cell, home, and work), email address, and home address will be obtained at the time of enrollment.

Data collection at the time of the procedure will be done either using a paper case report form (CRF) or directly into RedCap using a private bedside tablet. Prior to use, the paper CRF will be kept in the study packets. When used, paper data collection forms will have the subject's study number only. After the CRF is completed, it will be placed in a secure locked box in the ED until research personnel can transfer the CRF to a secure locked cabinet in the research office.

Research personnel will note the reason for the device's removal when it occurs. Study participants will be followed in their respective inpatient units. Study personnel will visit subjects daily to determine if the study IVs inserted in the ED are still in place. (Note. If study personnel are not available because of weekends or holidays, the study personnel will do their best to capture this information the next day possible.) Investigators will also document whether vasopressor medications have been administered through the IV and, if available, for what duration. Investigators will also make note of any nursing assessment of the lines for function and/or complication (e.g., blood return, erythema, oozing/bleeding, hematoma, concern for infection, infiltration, extravasation, need for treatment for vesicant infiltration, limb ischemia/tissue necrosis, presence of thrombus). Study staff may note what type of substances are being infused through the catheter (e.g., blood transfusion). Arm circumference will not be measured after original placement. From the participant's EHR, the investigators will also capture each additional IV that is placed and the associated billing from that procedure.

Each subject will remain in the study for 1-month following study VAD removal. If the subject remains hospitalized after the study device is removed, research staff will perform a clinical assessment by visiting the subject for 2 days following removal followed by a chart review at 1-week and 28-days post study device removal. If the subject is discharged within 28-days of study device removal, research staff will contact participants by phone 1-month from the date of discharge to ask about complications related to the device insertion and perform a chart review. If the study device remains until the date of discharge or the subject is discharged to home with the device in place, the subject will be called 1-month after discharge to ascertain outcomes.

Sample Size Calculation and Data analysis The investigators estimate, given our resources and ED census of eligible patients, that the investigators can recruit at least 70 and a maximum of 120 subjects per group over 24 months. The investigators are basing our sample size assuming the investigators can enroll the maximum number of subjects, which is 120 subjects in each arm, or 240. The investigators also plan to add an additional 30 subjects to account for potential missing primary outcome data or withdrawals. Therefore, our total sample size is a maximum of 270 subjects.

The investigators plan to compare long PIVs and MCs via three different parameters. For a 0.05 level of alpha and two-sided tests of hypotheses, below are our estimates of power to detect effect sizes based on the respective methods of analyses given our subjects recruitment capabilities:

1. Comparison of rates of completion of care by VAD (primary outcome) Hypothesis: The cumulative hazard of failure of midline catheters in the first 5 days is significantly lower than standard catheters over the same period. Assuming a 20% cumulative survival of the long PIVs by day 5, a sample of 120 subjects in each group will provide 80% power to differentiate from midline catheters with survival probability of 35.2% or greater. However, with 70 subjects in each group, to get 80% power the midline catheter survival probability would need to be at least 41%. In our opinion, both of these differences in survival probabilities (35.2% and 41%) are clinically meaningful and would lead to a change in clinical practice.
2. Comparison of proportions of failures at a fixed time after insertion of catheter.

   Hypothesis: The proportion of subjects whose catheters would fail by 5 days will be significantly higher for long PIVs as compared to midline catheters. Assuming 80% of long PIVs fail by day 5, a sample of 120 subjects in each group will give us 80% power to differentiate from midline catheters with an expected failure rate of 63.8% or lower. However, sample of 70 subjects in each group would provide 80% power to differentiate from midline catheters with an expected failure rate of 58% or lower.
3. Comparisons of mean time to failures of the two catheter types Hypothesis: The mean days to failure/removal will be 1.5 days longer for midline catheters as compared to standard catheters. A sample size of 113 subjects in each group will provide us 80% power to detect a minimum difference in mean catheter days of 1.5 days, assuming a common standard deviation as large as 4 days. A sample of 120 subjects would increase the power to 82.5%. However, a sample of 70 subjects in each group would have 80% power detect a minimum difference of 2 days.

DATA ANALYSIS

Data will be entered into a REDCap™ data collection form which is encrypted and password protected. Subjects will be analyzed using an intention to treat analysis, although the investigators will also perform a per protocol analysis as well for the final study results.

The primary outcome measure is survival of each venous access device. Secondary outcomes include complications, adverse events, and subject satisfaction, and will be determined based on review of the clinical record and subject responses to a questionnaire. Kaplan-Meier curves, log-rank test, Cox-proportional hazard ratio, t-tests for difference in proportions, and means will be used for analyses where appropriate.

Aim 1: Catheter dwell time Overall catheter survival will be determined by how long the catheter is in place and functional. The primary outcome will be to determine if the VAD remains inserted and function through completion of care, defined as a) present until time of discharge or b) present until the need for vascular access is completed. The investigators will report data based on a Kaplan Meier curve to display catheter survival. The investigators will also report the proportion of each type of catheter that is in place and functional at 3 days and 5 days post placement and the median dwell times. Dr. Ashar Ata, a biostatistician in the Department of Emergency Medicine will perform the statistical analysis of the data.

Aim 2: Complication rates The investigators will measure and compare the proportion of complications in each study arm. The investigators will record the qualitative type of complication (if any) experienced in each study arm for potential comparison of complication rates by complication type.

Aim 3: To determine subject experience, satisfaction, and preference; provider perceptions and cognitive load; and operational characteristics for each device placement.

The investigators will compare subject questionnaire responses, provider (proceduralists) questionnaire responses, and operational characteristics based on descriptive statistics, chi-square tests, or t tests as appropriate. The investigators will compare the time to placement (based upon time-motion measurements) in each study arm.

The investigators will perform a pilot analysis at the end of the first week of the 4th subject's enrollment. This planned analysis will be performed with the intention of optimizing the flow of the protocol and adequate data collecting. The interventions and outcomes will not be adjusted as a part of this planned review. The investigators will review these 4 subjects to review protocol flow and data collection fields. Amendments to the protocol or data collection form are required, will be submitted to the IRB prior to enrolling the 5th subject.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and older) patients presenting to the AMC ED with difficult IV access defined as any of the following:

  * Two failed attempts at landmark based IV or US-guided peripheral vascular access by qualified ED staff
  * Self-reported history of difficult IV access and one of the following:

    * History of requiring 2 or more IV attempts on a previous visit (either self-reported or documented in the electronic medical record)
    * Previous requirement for a rescue device after failed IV access attempt. These devices are as follows:
* US guided PIV
* Midline catheter
* Peripherally inserted central catheter
* Central venous catheter
* Intraosseous catheter
* History of or active comorbid disease state with known difficult IV access
* Prior or current implanted port device
* End stage renal disease with fistula
* Sickle cell disease
* History of or active intravenous drug use

Exclusion Criteria:

* Patients under the age of 18
* Known Prisoners
* Non-English-speaking patients
* Patients in whom the device cannot be stabilized due to tissue or treatments in bilateral extremities or available extremity (burns, complex humeral fractures, dialysis fistulas etc.)
* Patients lacking capacity to consent
* Patients unable to sign written consent
* Patients without identifiable target veins by ultrasonography
* Known pregnant patients
* Previously enrolled in this study
* Previously withdrawn from this study
* Presented when no study IV proceduralists are available
* Patients in whom obtaining informed consent and being enrolled in the study would put them at risk for obtaining time sensitive medical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-10-21 (Estimated); Study Completion 2027-10-21 (Estimated)

PRIMARY OUTCOMES:
Completion of Care and catheter dwell time | From enrollment through time to vascular access device removal, up to 28 days
  Catheter dwell time until completion of care will be measured. Completion of care will be considered to be the time of insertion of the study VAD to either a) discharge from the hospital or b) a documented completion of need for IV therapy warranting removal of the study VAD. Overall catheter survival will be determined by how long the catheter is in place and functional. We will report data based on a Kaplan Meier curve to display catheter survival.

SECONDARY OUTCOMES:
Complication Rates | through study completion, an average of 2 months.
  We will measure and compare the proportion of complications in each study arm. We will record the qualitative type of complication (if any) experienced in each study arm for potential comparison of complication rates by complication type.
Patient experience, satisfaction, and preference | At the time of patient enrollment
  We will compare subject questionnaire responses, provider (proceduralists) questionnaire responses, and operational characteristics based on descriptive statistics, chi-square tests, or t tests as appropriate. This will be performed on a 10-point Likert scale, where higher scores are better outcomes.
Procedural Time | At the time of patient enrollment
  We will measure how long it takes to complete each procedure, including set up time.
3- and 5-day dwell time | From enrollment through time to vascular access device removal, up to 28 days
  We will also report the proportion of each type of catheter that is in place and functional at 3 days and 5 days post placement and the median dwell times.
Procdural Time | At enrollment through device insertion, up to 2 hours
  We will compare the time (in minutes) to device insertion (based upon time-motion measurements) in each study arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center Hospital, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
We may plan to use study as a foundation for future, multicenter prospective study

REFERENCES:
- [Result] Prasanna N, Yamane D, Haridasa N, Davison D, Sparks A, Hawkins K. Safety and efficacy of vasopressor administration through midline catheters. J Crit Care. 2021 Feb;61:1-4. doi: 10.1016/j.jcrc.2020.09.024. Epub 2020 Oct 2. PMID 33049486
- [Result] Tripathi S, Kumar S, Kaushik S. The Practice and Complications of Midline Catheters: A Systematic Review. Crit Care Med. 2021 Feb 1;49(2):e140-e150. doi: 10.1097/CCM.0000000000004764. PMID 33372744
- [Result] Bahl A, Hang B, Brackney A, Joseph S, Karabon P, Mohammad A, Nnanabu I, Shotkin P. Standard long IV catheters versus extended dwell catheters: A randomized comparison of ultrasound-guided catheter survival. Am J Emerg Med. 2019 Apr;37(4):715-721. doi: 10.1016/j.ajem.2018.07.031. Epub 2018 Jul 19. PMID 30037560
- [Result] Greenwald RA, Rheingold OJ, Chiprut RO, Rogers AI. Local gangrene: a complication of peripheral Pitressin therapy for bleeding esophageal varices. Gastroenterology. 1978 Apr;74(4):744-6. PMID 305380
- [Result] Anderson JR, Johnston GW. Development of cutaneous gangrene during continuous peripheral infusion of vasopressin. Br Med J (Clin Res Ed). 1983 Dec 3;287(6406):1657-8. doi: 10.1136/bmj.287.6406.1657. PMID 6416538
- [Result] Elia F, Ferrari G, Molino P, Converso M, De Filippi G, Milan A, Apra F. Standard-length catheters vs long catheters in ultrasound-guided peripheral vein cannulation. Am J Emerg Med. 2012 Jun;30(5):712-6. doi: 10.1016/j.ajem.2011.04.019. Epub 2011 Jun 23. PMID 21703801
- [Result] Bahl A, Hijazi M, Chen NW, Lachapelle-Clavette L, Price J. Ultralong Versus Standard Long Peripheral Intravenous Catheters: A Randomized Controlled Trial of Ultrasonographically Guided Catheter Survival. Ann Emerg Med. 2020 Aug;76(2):134-142. doi: 10.1016/j.annemergmed.2019.11.013. Epub 2020 Jan 16. PMID 31955940
- [Result] Keyes LE, Frazee BW, Snoey ER, Simon BC, Christy D. Ultrasound-guided brachial and basilic vein cannulation in emergency department patients with difficult intravenous access. Ann Emerg Med. 1999 Dec;34(6):711-4. doi: 10.1016/s0196-0644(99)70095-8. PMID 10577399